CLINICAL TRIAL: NCT01637155
Title: Study to Evaluate the Pharmacokinetics of Vitamin D (Cholecalciferol) in Patients Undergoing Obesity Surgery in a Deficit Situation and After Standardization
Acronym: PK-VIT-D
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PK-VIT-D
Record Dates: First submitted 2012-07-10; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Obesity; Gastric Bypass; Gastrectomy
Keywords: Cholecalciferol
MeSH Terms: conditions — Obesity | interventions — Cholecalciferol; Chocolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cholecalciferol (Experimental)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — One baseline oral dose of 50.000 UI to determine pharmacokinetics. After 28 days, patients take a period of 90 days of standardization of cholecalciferol based on baseline levels. After this period, patients receive a second oral dose of 50.000 UI to determine a second pharmacokinetics.
  Other Names: Oral Cholecalciferol for pharmacokinetics determination:; - VITAMIN D3 Kern Pharma mixed with chocolate or vanilla custard; Standarization cholecalciferol dose depends on baseline levels as indicated below:; - <10 2800 UI; - 10-15 2000 UI; - 15-20 1200 UI; - 20-30 1000 UI

SUMMARY:
Set the pattern of vitamin D supplementation in obese patients undergoing bariatric surgery in deficit of vitamin D.

Patients receive a single oral dose of vitamin D, during the 28 days will be done a kinetic curve. Then and over the next 3 months, levels are normalized. Once normalized, will be administered another single oral dose to a second pharmacokinetic evaluation.

DETAILED DESCRIPTION:
The study is conducted in obese patients undergoing bariatric surgery (for bypass or sleeve gastrectomy) in deficit of vitamin D.

Will include a total of 44 patients, 22 from each type of surgery. Patients receive a single oral dose of vitamin D of 50,000 IU. During the 28 days after administration of vitamin D will be done a kinetic curve determining plasma levels of vitamin D on 15 occasions. Then and over the next 3 months, levels are normalized by providing a daily oral dose for each patient. Once levels are normalized, will be administered another single oral dose of 50,000 IU vitamin D and proceed to a second pharmacokinetic evaluation determining plasma levels 15 times.

Patient follow up is approximately 36 weeks. Patients go to the screening visit, baseline visit and visits on days 1, 2, 3, 14 and 28 days after each pharmacokinetic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years old
* with bariatric surgery in the last 18 months (+/- 6 months)
* BMI: 25-33 kg/m2
* vitamin D3 (OK)<20ng/mL.
* Clinically stable, in the opinion of the investigator, at the time of inclusion
* Signed consent form

Exclusion Criteria:

* pregnancy, lactation or intention during the study period.
* menopause
* GOP, GPT>2 UNL
* glomerular filtration rate <60ml/min
* previous renal lithiasis
* any digestive disease to suggest malabsorption, granulomatous diseases, diabetic gastroenteropathy and taking medication likely to interfere with the absorption of vitamin D and bone metabolism such as corticosteroids and anticonvulsants
* taking medication that interferes with calcium metabolism.
* cholecalciferol hypersensitivity.
* other bariatric surgery (different of by-pass or tubular gastrectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)

PRIMARY OUTCOMES:
Comparison of pharmacokinetic parameters | 36 weeks
  Comparison of the pharmacokinetic parameters of vitamin D according to a non compartimental approach (AUC0-t, AUC0-∞, Cmax and t1/2) between a state of vitamin D and after normalization of the same.

SECONDARY OUTCOMES:
Comparison of the pharmacokinetic parameters between the two types of surgery | 36 weeks
  Comparison of the pharmacokinetic parameters of vitamin D according to a non-compartmental approach (AUC0-t, AUC0-∞, Cmax and t1 / 2) between the two types of surgery (bypass and sleeve gastrectomy)
Proportion of patients with secondary hyperparathyroidism in both surgeries. | 36 weeks
Change from baseline levels of urinary excretion of calcium in both surgeries | 36 weeks
Change from baseline levels of urinary excretion creatinine in both surgeries | 36 weeks
Change from baseline in both biochemistry surgery | 36 weeks
  Changes in total protein, albumin, phosphorus, magnesium and calcium will be analyzed.
Change from baseline alkaline phosphatase levels in both surgeries | 36 weeks
Change from baseline body fat distribution by DEXA | 36 weeks
Changes adherence in both surgeries | 36 weeks
Incidence of adverse and clinical laboratory events for each of the surgeries | 36 weeks
Proportion of patients with serious adverse events related to medication | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Violeta Moize, MD, Principal Investigator — Hospital Clinic i provincial de Barcelona
Locations (1):
- Hospital Clinic i Provincial Barcelona, Barcelona, Barcelona, Spain